CLINICAL TRIAL: NCT00280670
Title: CBT for Comorbid Anxiety Disorders in Children With Autism, Asperger Syndrome, or PDD-NOS
Acronym: BIACA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Jeffrey J. Wood, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R03MH075806-01 (NIH)
Record Dates: First submitted 2006-01-20; First posted 2006-01-23 (Estimated); Last update posted 2012-04-02 (Estimated); Status verified 2012-03

CONDITIONS: Autistic Disorder; Asperger Syndrome; Anxiety Disorders
MeSH Terms: conditions — Autistic Disorder; Asperger Syndrome; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Behavioral Therapy (Experimental)
  Interventions: Behavioral: Cognitive-behavioral therapy
- Waitlist (No Intervention)

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy — Cognitive behavioral therapy for children with autism and anxiety.
  Arms: Cognitive Behavioral Therapy

SUMMARY:
This study is designed to examine the efficacy of a cognitive behavioral therapy (CBT) program for treating anxiety symptoms, social problems, and adaptive behavior deficits in children with autism spectrum disorders.

DETAILED DESCRIPTION:
Anxiety disorders are commonly diagnosed in children with autism, Asperger syndrome (AS), and pervasive developmental disorder not otherwise specified (PDD-NOS). Anxiety disorders contribute to children's functional impairment over and above the functional deficits attributable to autism, AS, and PDD-NOS. Thus, investigators have called for the development of anxiety treatments for this population (Attwood, 2003). Cognitive behavioral therapy (CBT) has been found to be efficacious for anxiety disorders in typically developing children. This pilot study will advance the field by providing an estimate of the treatment effects of CBT for anxiety disorders among children with autism, AS, or PDD-NOS. The sample will include 20 children aged 7-11 years with autism, AS, or PDD-NOS and a comorbid anxiety disorder. Children will be randomly assigned to immediate treatment or a 3-month waitlist. The manualized CBT program includes traditional anxiety treatment components including coping skills training (e.g., cognitive restructuring), in vivo exposure, operant procedures, and parent training. Additional treatment components have been added to enhance intervention response in children with AS or PDD-NOS, including emotion education, social skills/friendship skills training, and peer tutoring/mentoring modules. Trained graduate students with expertise in CBT and developmental disabilities will serve as therapists. Treatment fidelity will be checked using a session-by-session adherence checklist. Treatment acceptability and consumer satisfaction will be assessed at posttreatment, providing guidance on the extent to which the manual will need to be revised. Multiple measures of children's anxiety, including a structured diagnostic interview administered by an independent evaluator, will comprise the primary outcomes. Children's social functioning, adaptive behavior, and service use will also be assessed to determine if CBT can affect relevant distal outcomes. By comparing outcomes for children in the immediate treatment group versus those in the waitlist group, we will estimate effect sizes of CBT for this population. Subsequently, power analyses will be conducted in planning for a larger clinical trial. This study could contribute to public health efforts to address the mental health needs of the rising number of children diagnosed with autism-spectrum disorders. If CBT is found to be efficacious, it will be the first evidence-based psychological treatment to be successfully adapted for children with autism, AS, and PDD-NOS.

ELIGIBILITY:
Inclusion Criteria:

* 7 - 11 years of age
* Meet research criteria for a diagnosis of Asperger Syndrome or PDD-NOS
* Meet DSM-IV criteria for one of the following anxiety disorders: Separation Anxiety Disorder, Social Phobia, Obsessive-Compulsive Disorder
* If taking medication, have maintained a stable dose for 1 month prior to baseline assessment

Exclusion Criteria:

* Child has an IQ of less than 70
* Begin taking new medication(s) or current medication dose changes either (1) less than 1 month prior to baseline assessment, or (2) during the study period
* For any reason the child or parents appear unable to participate in the treatment program

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2005-01; Primary Completion 2008-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Score on anxiety diagnostic interview after treatment or waitlist | post-treatment
Score on anxiety rating scale after treatment or waitlist | post-treatment

SECONDARY OUTCOMES:
Score on daily living skills rating scale after treatment or waitlist | post-treatment
Score on children's social functioning and service use after treatment or waitlist | post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J Wood, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Derived] Wood JJ, Drahota A, Sze K, Har K, Chiu A, Langer DA. Cognitive behavioral therapy for anxiety in children with autism spectrum disorders: a randomized, controlled trial. J Child Psychol Psychiatry. 2009 Mar;50(3):224-34. doi: 10.1111/j.1469-7610.2008.01948.x. PMID 19309326
- See also: UCLA Center for Autism Research and Treatment — http://www.autism.ucla.edu